CLINICAL TRIAL: NCT05922449
Title: Using Thoracic Paravertebral Block for Perioperative Lung Preservation During VATS Pulmonary Surgery: A Dual Center Randomized Controlled Trial
Brief Title: Using Thoracic Paravertebral Block for Perioperative Lung Preservation During VATS Pulmonary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TREC2023-KY020
Record Dates: First submitted 2023-06-01; First posted 2023-06-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pulmonary Complications
Keywords: Postoperative pulmonary complications; Thoracic paravertebral block; Postoperative analgesia; Video-Assisted Thoracoscopic Surgery

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Packet information is hidden in serially numbered, sealed and opaque envelopes for allocation hiding.
  Due to the different anesthesia methods implemented in this study, the operators cannot achieve the blind method. The outcome assessor and data statisticians are blinded to the group assignment. If a major adverse event occurs during perioperative period that poses a serious threat to the safety of the subject and the anesthesiologist or attending physician deems it necessary to know the subject's grouping, an authorized blind person may open an emergency blind letter, record the time, cause and name of the blind person, and immediately report it to the supervisory board.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block group (PV group) (Experimental): This group of patients will undergo ultrasound-guided thoracic paravertebral nerve block in T4 and T7 thoracic paravertebral spaces before general anesthesia.
  Interventions: Procedure: Thoracic Paravertebral Block
- Control group (C group) (No Intervention): This group of patients did not undergo any nerve block procedures before general anesthesia.

INTERVENTIONS:
Procedure: Thoracic Paravertebral Block — Patients randomly assigned to PV group will be placed in lateral position, and punctured using the out of plane technique guided by ultrasound (Shenzhen Huasheng Navi low-frequency convex array probe). 15 ml of 0.5% ropivacaine was administered to the T4 and T7 thoracic paravertebral spaces respectively, for a total of 30 ml. After injection, the pleura of the punctured segment and adjacent segments could be obviously moved down. Upon successful puncture, the patient was transferred to the supine position. After 5, 10, and 15 minutes, the range of sensory blockage was tested at T3~T8 to cover the surgical area.
  Arms: Paravertebral block group (PV group)

SUMMARY:
Background: Postoperative pulmonary complications (PPCs) may extend the length of stay of patients and even increase perioperative mortality after video-assisted thoracoscopic (VATS) pulmonary surgery. Thoracic paravertebral block (TPVB) can provide effective analgesia after VATS, however little is known about the effect of TPVB on PPCs. This study aims to determine whether TPVB combined with general anesthesia results in reducing PPCs and achieve perioperative lung protection in VATS pulmonary surgery compared with simple general anesthesia.

Methods: A total of 302 patients undergoing VATS lobectomy/segmentectomy will be randomly divided into two groups: Paravertebral block group (PV group) and Control group (C group). Patients of PV group will receive thoracic paravertebral block: 15 ml of 0.5% ropivacaine will be administered to the T4 and T7 thoracic paravertebral spaces respectively before general anesthesia. Patients of C group will not undergo intervention. Both groups of patients adopted protective ventilation strategy during operation. Perioperative protective mechanical ventilation and standard fluid management will be applied in both groups. Patient controlled intravenous analgesia was used for postoperative analgesia. The primary endpoint is the composite outcome of PPCs within 7 days after surgery. Secondary end points include blood gas analysis, postoperative lung ultrasound score, NRS score, QoR-15 score, hospitalization related indicators and long-term prognosis indicators.

DETAILED DESCRIPTION:
Surgical resection is still the go-to treatment for lung cancer, which is the leading cause of cancer death As a minimally invasive operation, video-assisted thoracoscopic surgery (VATS) has significantly reduced surgical trauma and systemic inflammation, and has become the standard treatment method for lung cancer.

Postoperative pulmonary complications (PPCs) are one of the most common complications after thoracoscopic lung cancer surgery, with an incidence of 40.8%. PPCs increase hospitalization time, hospitalization cost, and perioperative mortality, and affect the treatment effect and utilization of medical resources. One of the most pressing clinical issues is how to lower the prevalence of PPCs. Previous research has shown that lung protective ventilation strategies, including low tidal volume, positive end expiratory pressure (PEEP), low inhalation oxygen concentration, etc., have a good prognosis in patients with lung injury, but they may not fully prevent acute lung injury caused by one-lung ventilation (OLV) during VATS.

The incidence of pain 24 hours after VATS was 38%, and the incidence of chronic pain 6 months after VATS was 25%. Poor postoperative analgesia will affect postoperative recovery, which may raise the risk of pulmonary complications due to insufficient respiratory function and weak sputum excretion. Thus, it is crucial to effectively control acute discomfort following VATS.

Ultrasound guided thoracic paravertebral block (TPVB) is a commonly used regional block technique in thoracic surgery. Local anesthetics can be injected into the paravertebral space to block the ipsilateral sympathetic and somatosensory nerves. TPVB combined with general anesthesia (GA) can reduce the pain after VATS, decreases the expression of matrix metalloproteinase-9, reduce the inflammatory reaction after thoracic surgery, improve the postoperative survival rate by blocking the unilateral sympathetic nerve, improve the postoperative rehabilitation of patients after VATS lung cancer radical surgery, and reduce the postoperative tumor recurrence. According to a recent retrospective propensity matching analysis, TPVB and GA together were linked to a decreased incidence of PPCs (29.8% vs. 34.2%). However, a prospective study on the effects of GA combined with GA alone vs GA coupled with TPVB on PPCs following VATS pulmonary surgery has not been retrieved.

The aim of this study is designed to explore whether general anesthesia combined with thoracic paravertebral block can reduce atelectasis, lung inflammation, and lung injury compared to general anesthesia during VATS pulmonary surgery, thereby reducing the incidence of postoperative pulmonary complications, achieving lung protection, and improving long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective VATS lobectomy/segmentectomy had an expected operation duration (from skin incision to suture) greater than 1h
* Age>18
* American society of Anesthesiologists (ASA) physical status classification system: I - III

Exclusion Criteria:

* Patients with acute or chronic respiratory failure, chronic obstructive pulmonary disease (GOLD) grade ≥ Grade III, poorly controlled asthma or acute respiratory distress syndrome (ARDS, according to the new definition of ARDS at the 2011 Berlin Conference)
* Patients with severe cardiovascular complications (defined as New York Heart Association (NYHA) Grade IV, acute coronary syndrome, or persistent ventricular tachycardia)
* Patients who had a history of ipsilateral thoracotomy or had a history of mechanical ventilation within 4 weeks
* Patients with contraindications to TPVB (coagulation dysfunction, anticoagulation or antiplatelet therapy, skin ulcer infection, local anesthetic allergy, Spinal deformity, etc.)
* Patients with trachea malformation or tracheotomy
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The incidence of the composite of postoperative pulmonary complications (PPCs) within 7 days after surgery | Within the first 7 days after operation
  Unit: %; This value is a percentage. Patients with at least one complication were considered eligible for the primary end points.
  Postoperative pulmonary complications include pneumonia; aspiration pneumonitis; atelectasis; respiratory failure; bronchospasm; pulmonary congestion; pleural effusion; pneumothorax.

SECONDARY OUTCOMES:
Arterial partial pressure of oxygen (PaO2) | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: mmHg
Arterial carbon dioxide pressure (PaCO2) | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: mmHg
Oxygenation index (OI) | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  OI =PaO2/Inspired oxygen fraction (FiO2), Unit: mmHg
Arterial blood pH | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unitless
Concentration of arterial blood lactate | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: mmol/L
Heart rate | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: beats per minute
Invasive arterial blood pressure | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: mmHg
Transcutaneous oxygen saturation (SpO2) | Preoperative; one-lung ventilation (OLV) for 30 minutes; 5 minutes after the end of one lung ventilation; 30 minutes after entering the postoperative pulmonary complications (PACU)
  Unit: %; This value is a percentage
Lung Ultrasound Score (LUS) | Preoperative; Postoperative day1; Postoperative day 2
  Unit: point Operation method: Each side of the chest of the patient was divided into six regions with the front axillary line, the posterior axillary line, and the nipple line as the boundary. Use the ultrasonic probe to scan each area from right to left, from top to bottom, and from front to back.
  LUS score = sum of all 12 regions, Min = 0; Max = 36. The higher the score, the worse the degree of ventilation is considered.
  Score according to the number of B lines in the LUS image of each area. 0: B lines ≤ 2; 1 point: > 2 well-spaced B-lines; 2 points: Multiple coalescent B lines; 3 points: white lung (lung consolidation).
Numerical rating scale (NRS) | Preoperative; Postoperative day1; Postoperative day 2; 1 and 3 months after operation
  Unit: point, including chest NRS score for rest and cough. Participants were asked to rate their average pain intensity for rest and cough by selecting a single number from 0 to 10. The end-point descriptors for the NRS was "No pain"(0) to "The most intense pain imaginable" (10). The higher the score, the more severe the pain situation.
Patient's postoperative consumption of sufentanil | Within 48 hours after operation
  Provided through patient controlled intravenous analgesia (PCIA) equipment; Unit: mcg.
The incidence of opioid-related adverse effects | Within 48 hours after operation
  Unit: %; This value is a percentage. Opioid-related adverse effects include nausea, vomiting, dizziness, pruritus.
Quality of recovery with the 15-item (QoR-15) | Preoperative; Postoperative day1; Postoperative day 2; 1 and 3 months after operation
  Unit: point. QoR-15 is a global measure of recovery after surgery that evaluates five dimensions of recovery: physical comfort (5 items), physical independence (2 items), emotional state (4 items), psychological support (2 items), and pain (2 items). Each item is rated on an 11- point scale based on its frequency on the questionnaire (greater score at greater frequency for positive items and less frequency for negative items). The total score ranged from 0 (poorest recovery quality) to 150 (best recovery quality).
The incidence of various postoperative pulmonary complications | Within the first 7 days after surgery; 1 and 3 months after operation
  Unit: %; This value is a percentage. Postoperative pulmonary complications include pneumonia; aspiration pneumonitis; atelectasis; respiratory failure; bronchospasm; pulmonary congestion; pleural effusion; pneumothorax.
The incidence of various postoperative extrapulmonary complications | Within the first 7 days after surgery; 1 and 3 months after operation
  Unit: %; This value is a percentage. Postoperative pulmonary complications include arrhythmia; cardiovascular complications (arrhythmias, acute coronary syndrome, mycardial infarction, acute congestive heart failure); cerebrovascular complications (cerebral infarction, cerebral hemorrhage); postoperative cognitive dysfunction (POCD); postoperative renal complications; shock; postoperative extrapulmonary infection.
Postoperative mortality rate | 1 and 3 months after operation
  Unit: %; This value is a percentage.
Unplanned ICU hospitalization rate | 1 months after operation
  Unit: %; This value is a percentage.
Unplanned ICU hospitalization duration | 1 months after operation
  Unit: Hour.
Postoperative length of stay | 1 months after operation
  Unit: Day. from date of operation till date of discharge
Hospitalization expense | 1 months after operation
  Unit: CNY.

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Study Director — Beijing Tongren Hospital
Locations (2):
- China (2):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing tongren Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Result] Falcoz PE, Puyraveau M, Thomas PA, Decaluwe H, Hurtgen M, Petersen RH, Hansen H, Brunelli A; ESTS Database Committee and ESTS Minimally Invasive Interest Group. Video-assisted thoracoscopic surgery versus open lobectomy for primary non-small-cell lung cancer: a propensity-matched analysis of outcome from the European Society of Thoracic Surgeon database. Eur J Cardiothorac Surg. 2016 Feb;49(2):602-9. doi: 10.1093/ejcts/ezv154. Epub 2015 Apr 26. PMID 25913824
- [Result] Lohser J, Slinger P. Lung Injury After One-Lung Ventilation: A Review of the Pathophysiologic Mechanisms Affecting the Ventilated and the Collapsed Lung. Anesth Analg. 2015 Aug;121(2):302-18. doi: 10.1213/ANE.0000000000000808. PMID 26197368
- [Result] Colquhoun DA, Leis AM, Shanks AM, Mathis MR, Naik BI, Durieux ME, Kheterpal S, Pace NL, Popescu WM, Schonberger RB, Kozower BD, Walters DM, Blasberg JD, Chang AC, Aziz MF, Harukuni I, Tieu BH, Blank RS. A Lower Tidal Volume Regimen during One-lung Ventilation for Lung Resection Surgery Is Not Associated with Reduced Postoperative Pulmonary Complications. Anesthesiology. 2021 Apr 1;134(4):562-576. doi: 10.1097/ALN.0000000000003729. PMID 33635945
- [Result] Lederman D, Easwar J, Feldman J, Shapiro V. Anesthetic considerations for lung resection: preoperative assessment, intraoperative challenges and postoperative analgesia. Ann Transl Med. 2019 Aug;7(15):356. doi: 10.21037/atm.2019.03.67. PMID 31516902
- [Result] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Result] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Result] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Result] Tong C, Zhu H, Li B, Wu J, Xu M. Impact of paravertebral blockade use in geriatric patients undergoing thoracic surgery on postoperative adverse outcomes. J Thorac Dis. 2019 Dec;11(12):5169-5176. doi: 10.21037/jtd.2019.12.13. PMID 32030234
- [Result] Ben Aziz M, Mukhdomi J. Thoracic Paravertebral Block. 2023 Feb 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK570560/ PMID 34033322
- [Result] Kang K, Meng X, Li B, Yuan J, Tian E, Zhang J, Zhang W. Effect of thoracic paravertebral nerve block on the early postoperative rehabilitation in patients undergoing thoracoscopic radical lung cancer surgery. World J Surg Oncol. 2020 Nov 12;18(1):298. doi: 10.1186/s12957-020-02071-8. PMID 33183325
- [Result] Chu H, Dong H, Wang Y, Niu Z. Effects of ultrasound-guided paravertebral block on MMP-9 and postoperative pain in patients undergoing VATS lobectomy: a randomized, controlled clinical trial. BMC Anesthesiol. 2020 Mar 6;20(1):59. doi: 10.1186/s12871-020-00976-1. PMID 32143570
- [Result] Tong C, Zheng J, Wu J. The effects of paravertebral blockade usage on pulmonary complications, atrial fibrillation and length of hospital stay following thoracoscopic lung cancer surgery. J Clin Anesth. 2022 Aug;79:110770. doi: 10.1016/j.jclinane.2022.110770. Epub 2022 Mar 22. PMID 35334289
- [Result] Kimura A, Suehiro K, Juri T, Fujimoto Y, Yoshida H, Tanaka K, Mori T, Nishikawa K. Hemodynamic Changes via the Lung Recruitment Maneuver Can Predict Fluid Responsiveness in Stroke Volume and Arterial Pressure During One-Lung Ventilation. Anesth Analg. 2021 Jul 1;133(1):44-52. doi: 10.1213/ANE.0000000000005375. PMID 33687175
- [Result] de la Gala F, Pineiro P, Reyes A, Vara E, Olmedilla L, Cruz P, Garutti I. Postoperative pulmonary complications, pulmonary and systemic inflammatory responses after lung resection surgery with prolonged one-lung ventilation. Randomized controlled trial comparing intravenous and inhalational anaesthesia. Br J Anaesth. 2017 Oct 1;119(4):655-663. doi: 10.1093/bja/aex230. PMID 29121283
- [Result] Brassard CL, Lohser J, Donati F, Bussieres JS. Step-by-step clinical management of one-lung ventilation: continuing professional development. Can J Anaesth. 2014 Dec;61(12):1103-21. doi: 10.1007/s12630-014-0246-2. Epub 2014 Nov 12. English, French. PMID 25389025
- [Result] Kaufmann KB, Loop T, Heinrich S; Working Group of the German Thorax Registry. Risk factors for post-operative pulmonary complications in lung cancer patients after video-assisted thoracoscopic lung resection: Results of the German Thorax Registry. Acta Anaesthesiol Scand. 2019 Sep;63(8):1009-1018. doi: 10.1111/aas.13388. Epub 2019 May 29. PMID 31144301
- [Result] Wu Z, Fang S, Wang Q, Wu C, Zhan T, Wu M. Patient-Controlled Paravertebral Block for Video-Assisted Thoracic Surgery: A Randomized Trial. Ann Thorac Surg. 2018 Sep;106(3):888-894. doi: 10.1016/j.athoracsur.2018.04.036. Epub 2018 May 12. PMID 29763594
- [Result] Jung DM, Ahn HJ, Jung SH, Yang M, Kim JA, Shin SM, Jeon S. Apneic oxygen insufflation decreases the incidence of hypoxemia during one-lung ventilation in open and thoracoscopic pulmonary lobectomy: A randomized controlled trial. J Thorac Cardiovasc Surg. 2017 Jul;154(1):360-366. doi: 10.1016/j.jtcvs.2017.02.054. Epub 2017 Mar 10. PMID 28412111
- [Result] Wang ML, Hung MH, Chen JS, Hsu HH, Cheng YJ. Nasal high-flow oxygen therapy improves arterial oxygenation during one-lung ventilation in non-intubated thoracoscopic surgery. Eur J Cardiothorac Surg. 2018 May 1;53(5):1001-1006. doi: 10.1093/ejcts/ezx450. PMID 29253106
- [Result] Li XF, Hu JR, Wu Y, Chen Y, Zhang MQ, Yu H. Comparative Effect of Propofol and Volatile Anesthetics on Postoperative Pulmonary Complications After Lung Resection Surgery: A Randomized Clinical Trial. Anesth Analg. 2021 Oct 1;133(4):949-957. doi: 10.1213/ANE.0000000000005334. PMID 33410611
- [Result] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Result] El-Tahan MR. Role of Thoracic Epidural Analgesia for Thoracic Surgery and Its Perioperative Effects. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1417-1426. doi: 10.1053/j.jvca.2016.09.010. Epub 2016 Sep 13. No abstract available. PMID 27955978
- [Result] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Result] Licker MJ, Widikker I, Robert J, Frey JG, Spiliopoulos A, Ellenberger C, Schweizer A, Tschopp JM. Operative mortality and respiratory complications after lung resection for cancer: impact of chronic obstructive pulmonary disease and time trends. Ann Thorac Surg. 2006 May;81(5):1830-7. doi: 10.1016/j.athoracsur.2005.11.048. PMID 16631680
- [Result] Liang XL, An R, Chen Q, Liu HL. The Analgesic Effects of Thoracic Paravertebral Block versus Thoracic Epidural Anesthesia After Thoracoscopic Surgery: A Meta-Analysis. J Pain Res. 2021 Mar 26;14:815-825. doi: 10.2147/JPR.S299595. eCollection 2021. PMID 33814927
- [Result] Casati A, Alessandrini P, Nuzzi M, Tosi M, Iotti E, Ampollini L, Bobbio A, Rossini E, Fanelli G. A prospective, randomized, blinded comparison between continuous thoracic paravertebral and epidural infusion of 0.2% ropivacaine after lung resection surgery. Eur J Anaesthesiol. 2006 Dec;23(12):999-1004. doi: 10.1017/S0265021506001104. Epub 2006 Jul 7. PMID 16824243
- [Derived] Zhu J, Wei B, Wu L, Li H, Zhang Y, Lu J, Su S, Xi C, Liu W, Wang G. Thoracic paravertebral block for perioperative lung preservation during VATS pulmonary surgery: study protocol of a randomized clinical trial. Trials. 2024 Jan 22;25(1):74. doi: 10.1186/s13063-023-07826-8. PMID 38254233

DOCUMENTS (1):
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT05922449/ICF_000.pdf